CLINICAL TRIAL: NCT03372733
Title: Effect of Dietary Omega-7 Palmitoleic Acid-Rich Oil on Lipoprotein Metabolism and Satiety in Adults
Brief Title: Dietary Omega-7 Palmitoleic Acid-Rich Oil on Lipoprotein Metabolism and Satiety in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 180019; 18-H-0019
Record Dates: First submitted 2017-12-13; First posted 2017-12-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09-22

CONDITIONS: Cardiovascular Disease
Keywords: Omega-7; Palmitoleic Acid; Monounsaturated Fatty Acids; Lipoproteins; Satiety
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects randomized to the control olive oil arm will take the equivalent to 3g of control /day in two divided doses (4 capsules a day) for 8 +/- 2weeks and cross-over to the palmitoleate-rich oil
  Interventions: Drug: control olive oil (COO)
- Group 2 (Experimental): Subjects randomized to the control olive oil arm will take the equivalent to 3g of control /day in two divided doses (4 capsules a day) for 8 +/- 2 weeks and cross-over to the palmitoleate-rich oil arm will take the equivalent to 3g of control /day in two divided doses (4 capsules a day) for 8 +/- 2 weeks and cross-over to the control olive oil
  Interventions: Drug: palmitoleate-rich oil (PLO)

INTERVENTIONS:
Drug: control olive oil (COO) — 2 capsules, 2 times a day after meals in a total of 4 capsules a day
  Arms: Group 1
Drug: palmitoleate-rich oil (PLO) — 2 capsules, 2 times a day after meals in a total of 4 capsules a day
  Arms: Group 2

SUMMARY:
Background:

Omega-7 fatty acids are found in the oil extracted from certain fish and nuts like macadamia. Palmitoleic acid is one of the most common omega-7 fatty acids. Many studies suggest that this oil is good for heart health. Researchers want to find out more about these potential benefits.

Objective:

To study how oil enriched with palmitoleic acid (Omega-7 oil) affects metabolism.

Eligibility:

Healthy adults at least 18 years old with no known history of cardiovascular disease.

Subjects not allergic to fish oil and fish products

Females that are not pregnant and are not planning a pregnancy during the length of the study

Design:

Participants will be screened with questions about their health, medical history, and medicines they take.

Participants will have 4 visits over 24 weeks. The visits may include:

* Blood drawn from a vein in the arm by a needle stick. Sometimes participants will have to fast before the blood draw.
* Vital signs (blood pressure, heart rate, and temperature) taken
* Body mass index measured
* Cardio-Ankle Vascular Index test may be performed. The stiffness of the participant s arteries will be measured by reading blood pressure in the arms and legs and monitoring the heart.
* Optional stool samples
* Pregnancy test
* A short review of participants physical activity and diet
* A supply of dietary supplements to take between visits. Participants will take 4 gel capsules a day.

Participants will keep a food and exercise journal

Compensation will be provided to subjects that complete the study

Check your eligibility for this study by clicking here: https://www.surveymonkey.com/r/DietaryOmega

DETAILED DESCRIPTION:
Serum cholesterol is transported by lipoproteins, such as VLDL, LDL, and HDL, which vary in their relationship to cardiovascular disease risk. LDL, for example, is proatherogenic, whereas HDL is cardio-protective. Palmitoleic acid (cis-C16:1 n-7), an omega-7 fatty acid with 16 carbons in length with a single double bound in the n-7 position, have been shown in mice and human to decrease proatherogenic lipoproteins, such as LDL, and reduce cardiovascular risk factors. This study will test the hypothesis that palmitoleate supplementation in humans will favorably alter the lipoprotein lipid profile in regard to cardiovascular disease risk. We will also assess other parameters related to lipoprotein composition and function, as well as other biomarkers related to coagulation and inflammation, which have previously been shown to be possibly affected by supplementation with omega-7 fatty acid. In addition, previous animal studies have indicated the palmitoleate induced satiety and suppressed body weight gain, possibly through enhancement of the release of satiety hormones. In this clinical trial, we therefore will also examine the effect of concentrated palmitoleate on satiety.

This clinical research project is designed as a pilot, randomized, double-blinded, crossover study that will investigate the effect of concentrated oil enriched with palmitoleate on lipoprotein metabolism and satiety. Subjects will either receive control olive oil enriched in oleic acid, a longer-chain monounsaturated fatty acid (cis-C18:1 n-9), or a concentrate oil supplement produced from pollock fish (rich in palmitoleate) for approximately 8-10 weeks, with a wash out period of 8-10 weeks between the two arms of the study. The study consists of 4 outpatient visits when laboratory or research samples will be performed. A 7-day food diary, pill count, and red cell membrane fatty acid levels will be monitored to assess compliance. The effect of the supplement on satiety will be assessed at each visit.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male and female participants 18 years of age or above.
* Subject must be healthy, with no known history of cardiovascular disease.
* Post-menopausal or women of childbearing potential must be non-lactating and using an effective form of birth control during the course of the study.
* Subject understands protocol and provides written, informed consent in addition to a willingness to comply with specified follow-up evaluations.
* Subjects with triglyceride levels above 100 mg/dL

EXCLUSION CRITERIA:

* Pregnancy, planned pregnancy (within the study period), or women currently breastfeeding.
* Subjects with allergy or known hypersensitivity to fish, omega-3-acid ethyl esters, omega-7 ethyl esters, other related drugs, or any component of study drugs
* Subjects with weight changes greater than 20% over the past 3 months.
* Subjects planning a significant change in diet or exercise levels.
* Subjects already consuming more than 2 g per day of MUFA, PUFA or other forms of fatty acid supplement if determined by the investigator as having a potential to interfere in the data quality or patient safety.
* Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, or other known conditions that could affect intestinal fat absorption.
* Subjects with any acute and life-threatening condition, such but not limited to as prior sudden cardiac arrest, acute myocardial infarction (last three months), stroke, embolism as per investigator assessment.
* Subjects taking supplements or medications that affect lipoproteins for at least the past 8 weeks, such as fish oil supplements, bile-acid sequestrants, plant sterol supplements, fibrates, statins, Niacin or PCSK9 inhibitors.
* Subjects being treated with tamoxifen, estrogens, or progestins that have not been stable for >4 weeks.
* Subjects initiating new medications or patients on multiple medications may also be excluded according to investigator discretion.
* Anticipated surgery during the study period.
* Liver enzymes (AST or ALT) levels above 3x upper limit of normal.
* Blood donation in the last 2 weeks or planned blood donation during the study.
* Subjects requiring regular transfusions for any reason.
* Subjects may also be excluded for any reason that may compromise their safety or the accuracy of research data or for not complying with protocol directions.
* Abnormal baseline laboratory values that are considered not clinically significant by the PI will not exclude the subject.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
changes in the LDL-cholesterol levels | 24 weeks
  The primary outcome measures of this study will be changes in the LDL-cholesterol levels. Secondary outcome measurements will be changes in TC, TG, HDL-C, and other lipids, lipoprotein particle number, HDL functional test (i.e. efflux study) composition and size, changes in appetite and/or satiety. Each subject will serve as their own control.

SECONDARY OUTCOMES:
changes in TC, TG, HDL-C, and other lipids, lipoprotein particle number, HDL functional test (i.e. efflux study) composition and size, changes in appetite and/or satiety | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0019.html
- See also: https://www.surveymonkey.com/r/DietaryOmega — https://www.surveymonkey.com/r/DietaryOmega